CLINICAL TRIAL: NCT04671823
Title: Changes in the Prevalence of Oncogenic HPV Types After Introduction of Prophylactic HPV Vaccine Program in Japan
Brief Title: Changes in the Prevalence of Oncogenic HPV Types
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Kanazawa Medical University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Toshiyuki Sasagawa, Professor, Kanazawa Medical University
Other Study IDs: I547
Record Dates: First submitted 2020-12-11; First posted 2020-12-17 (Actual); Last update posted 2020-12-23 (Actual); Status verified 2020-12

CONDITIONS: Papillomavirus Vaccines; Papillomavirus Infections
Keywords: Human Papillomavirus; Papillomavirus Vaccines; Papillomavirus Infections
MeSH Terms: conditions — Papillomavirus Infections

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — This study requires liquid based cytology samples (fixed cells).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In Japan, nationwide prophylactic HPV vaccination was implemented in 2010; a bivalent vaccine was given from 2010 to 2012, and a quadrivalent vaccine from 2012. However, the program essentially ceased in June 2013.

1. Our first objective is to examine the prevalence of 6, 11, 16, 18, 31, 33, 45, 52, and 58 targeted by the nonavalent HPV vaccine in young Japanese women, and identify changes in the prevalence of these HPV types from 2011- 2012 (as reported in JHERS-2016; Sasagawa T, J Med Virol, 2016) to the present time (2020-2021). Especially, the investigators will focus on the prevalence of HPV16 and 18 in women aged 21-26 years and compare these data to those of the previous study.
2. The investigators will assess the prevalence of HPV16 and 18 in women aged 16-18 years and compare these data to those of the HPV vaccine era (2010-2013).
3. The investigators will explore the prevalence of other high-risk HPV types (35, 39, 51, 56, 59, and 68), 11 probable high-risk types (26, 30,34, 53, 66, 67, 69, 70, 73, 82, and 85), and SILs in Japanese young women, since these types might be causative HPV types for cervical cancer in the future after world-wide HPV vaccination.

Currently, it is unclear whether HPV vaccination has reduced the prevalence of HPV16 and 18 in Japan. Our previous study (JHERS-2016; performed during 2011-2012; Sasagawa T, J Med Virol, 2016), the only population-based study on HPV prevalence at the commencement of prophylactic HPV vaccination in Japan, included prevalence data for HPV types 6, 11, 16, and 18 and the associated cervical abnormalities. The investigators hypothesize that the prevalence of HPV16 and 18 and the associated diseases (SILs) decreased significantly in women aged 21-26 years in the present, vaccinated group compared to that in similar aged women in 2010-2012 who were unvaccinated. In contrast, the prevalence of HPV and associated diseases may not differ in women aged 27-39 years between the two eras; such subjects may thus serve as a negative control group. Also, HPV prevalence may be higher in present women aged 16-18 years than in women in that age range during the vaccine era, as the former group have not been vaccinated against HPV.

The prevalence rates of the other unique high-risk types, namely HPV35, 39, 51, 56, 59, and 68, and probable high-risk types, HPV26, 20, 34, 53, 66, 67, 67, 70, 73, 82, and 85, are unlikely to have been affected by HPV vaccination. However, it is important to monitor the prevalences of these types and the associated SILs, because the types numbered above may become more significant as currently common HPV types are eliminated in the near future.

DETAILED DESCRIPTION:
Recently, HPV prevalence has decreased dramatically in the USA (Markowitz LE, Pediatrics, 2019). Surprisingly, the nonavalent vaccine optimally decreased the prevalence of the most common, high-risk HPV types and also reduced the incidence of premalignant cervical lesions (Mariani L, Int J Gynaecol Obstet, 2017). The data thus suggest that both the bivalent and quadrivalent HPV vaccines eliminate HPV16- and 18-associated cervical cancers.

Regrettably, in Japan, use of the bivalent and quadrivalent prophylactic HPV vaccines almost ceased, by government decree, in June 2013 (Hanley JBS, Lancet, 2015). However, about 70% of girls aged 13-18 years were immunized with these vaccines during 2010-2012. A small decrease in cervical intraepithelial neoplasia grade 3 (CIN3) has been observed in 20-year-old Japanese women who underwent HPV vaccination (Yagi A, Vaccine, 2019).The investigators recently found nationwide (unpublished) data suggesting that the incidence of condyloma has decreased in Japanese women aged in their early twenties, but has apparently increased in males. The decrease in women may be attributable to quadrivalent HPV vaccination, which protects against HPV6 and 11 infections. Further work is necessary, as statistical analysis is lacking, and the proportion of quadrivalent vaccinations among all vaccinations is unknown in Japan.

The investigators earlier reported a high prevalence of HPV infection and associated cervical abnormalities in 6,628 women aged 16-50 years. The work was performed from October 2011 to March 2012 and was reported in JHERS-2016 (Sasagawa T, J Med Virol, 2016). The investigators recorded demographic information including age, marital status, any history of or current sexually transmitted disease (STD), any cervical abnormalities, and any other gynecological problems. HPV genotyping (31 types) and the Pap test were performed for all subjects. This is the only study that has investigated HPV prevalence and cervical SILs in the general population. The information collected included sexual details and any history of HPV vaccination. Routine gynecological examination, the Pap test (employing liquid-based cytology [LBC]), and HPV genotyping of LBC samples were performed. These data allow us to compare the status of women in the vaccine and (present) no-vaccine era.

It is possible to essentially eliminate cervical cancer by implementation of nanovalent HPV vaccination and careful cancer screening (HPV testing). However, some specialists suggest that reductions in certain HPV types might induce increases in other HPV types that are not targeted by vaccination and not tested during cancer screening. Not only the existing 13 high-risk HPV types but also other HPV types considered to probably or possibly associated with high risk are found in some cervical cancer tissues (Halec G, J Pathology 2014). The investigators also found such HPV types in high-grade SILs, as reported in JHERS-2016 (Sasagawa T, J Med Virol, 2016) and a recent publication (Sakamoto J, Papillomavirus Res, 2019). Therefore, in the present project, the investigators will document the prevalence of all oncogenic HPV types, including the 13 recognized high-risk types and the probable high-risk types (HPV26, 30, 34, 53, 66, 67, 69, 70, 73, 82, and 85).

ELIGIBILITY:
Inclusion Criteria:

* Japanese women who seek cervical cancer screening or gynecological consultations
* Women with benign conditions
* 16-39 year-old
* Women must be sexually experienced, as defined by sexual contact (oral-genital or genital-genital) with at least one male or female partner.

Exclusion Criteria:

* Women with STDs
* Women with premalignant lesions of the cervicovaginal tract
* Women suffering from any cancer
* Women with any severe acute or chronic disease, and/or psychological problems

Ages: 16 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Japanese women (aged 16-39 years) who seek cervical cancer screening or gynecological consultations.
Sampling Method: Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2020-12 (Estimated); Primary Completion 2021-09-30 (Estimated); Study Completion 2022-03-31 (Estimated)

PRIMARY OUTCOMES:
The prevalence of HPV types targeted by the nonavalent HPV vaccine | 12 months
  Our first objective is to examine the prevalence of 6, 11, 16, 18, 31, 33, 45, 52, and 58 targeted by the nonavalent HPV vaccine in young Japanese women, and identify changes in the prevalence of these HPV types from 2011- 2012 (as reported in JHERS-2016; Sasagawa T, J Med Virol, 2016) to the present time (2020-2021). Especially, The investigators will focus on the prevalence of HPV16 and 18 in women aged 21-26 years and compare these data to those of the previous study.

REFERENCES:
- [Background] Sasagawa T, Maehama T, Ideta K, Irie T; Fujiko Itoh J-HERS Study Group. Population-based study for human papillomavirus (HPV) infection in young women in Japan: A multicenter study by the Japanese human papillomavirus disease education research survey group (J-HERS). J Med Virol. 2016 Feb;88(2):324-35. doi: 10.1002/jmv.24323. PMID 26147986